CLINICAL TRIAL: NCT06462690
Title: Effect of Care Provided with Skin Care Protocol on Skin Moisture Change, Dermatological Quality of Life and Patient Comfort in Elderly Patients: Randomized Controlled Study
Brief Title: Effect of Care Provided Through Skin Care Protocol on Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duygu AKÇA (Other)
Responsible Party: Sponsor-Investigator, Duygu AKÇA, Lecturer, Kafkas University
Organization: Kafkas University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022-TS-53
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Elderly Person; Comfort; Quality of Life; Skin Moisture; Skin

STUDY DESIGN:
Intervention Model Description: Experimental Group Control Group
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants were included in the study using the single-blind randomization method. Block randomization was used in the randomization process. Since the research is a thesis study, double blinding cannot be done because the researcher who collects the data and performs the application is the same. However, blinding will be applied wherever possible in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): After determining the patients who meet the inclusion criteria and are willing to participate in the study, their consent is obtained and the protocol is applied by the researcher one day before the application, when the patient feels ready, using the face-to-face interview technique (PIF), (DLQI), (GCS), (SEF). Pre-test data is collected by applying it. Vital signs are taken and recorded. Skin moisture is measured with the DMM device. Braden Risk Assessment Scale is applied. After the measurements, the patient is given care according to the care protocol, measurements are made again in between, and then (DLQI), (GCS) is applied, and the skin moisture and vital signs are measured, and the process is concluded.
  Interventions: Other: pre-mid-post test
- Control Group (No Intervention): After the patients who meet the inclusion criteria and are willing to participate in the study are determined, their consent will be obtained and pre-test data will be collected by applying face-to-face interview techniques (PIF), (DLQI), (GCS) at a time when the patient feels ready. Vital signs will be taken and recorded. Skin moisture measurement will be made with a DMM device. Braden Risk Assessment Scale will be applied. After the measurements, according to the care protocol, the patients will not be given care, they will receive routine care, then (DLQI), (GCS) will be applied, skin moisture and vital signs will be measured and the procedure will be terminated.

INTERVENTIONS:
Other: pre-mid-post test — (PIF) (DLQI) (GCS) Data Collection Forms Humidity measurement with DMM device
  Arms: Experimental Group

SUMMARY:
The rate of elderly population is increasing in the world. It is reported that the proportion of the world population over the age of 60 will increase to 22% by 2050. With advancing age, the skin is inevitably affected and becomes more vulnerable to possible damage. Additionally, as the skin ages, it undergoes many internal and external deteriorations. Intrinsic aging refers to biological changes that cannot be prevented to a large extent. External factors; exposure to conditions such as ultraviolet rays and radiation. In addition, in elderly individuals, conditions such as frequent washing, especially washing with harsh products, lack of hygiene, trauma, decreased peripheral satisfaction, immobility, incontinence, diabetes, vascular changes, malnutrition, use of multiple medications, depression, and dementia are among the situations that increase the risk of deterioration in skin health Hypotheses of the Research H0-1=The care given to elderly patients according to the protocol prepared has no effect on the moisture status of the skin.

H1-1= The care given to elderly patients according to the prepared protocol affects the moisture status of the skin.

H0-2== The care given to elderly patients with the prepared protocol has no effect on their dermatological lives.

H1-2== The care given to elderly patients with the prepared protocol has an impact on their dermatological lives.

H0-3= The care provided with the protocol prepared for elderly patients has no effect on general comfort.

H1-3= The care provided with the protocol prepared in elderly patients has an effect on general comfort.

DETAILED DESCRIPTION:
The rate of elderly population is increasing in the world. It is reported that the proportion of the world population over the age of 60 will increase to 22% by 2050. This aging of the population is one of the most important factors affecting the population demographic structure of all countries in the world. These demographic changes create many challenges in all healthcare systems and care settings around the world. Age-related morphological and functional changes affect the whole body, as well as negatively affecting the skin, which is the largest organ of the body. With advancing age, the skin is inevitably affected and becomes more vulnerable to possible damage. Additionally, as the skin ages, it undergoes many internal and external deteriorations. Intrinsic aging refers to biological changes that cannot be prevented to a large extent. External factors; exposure to conditions such as ultraviolet rays and radiation. In addition, in elderly individuals, conditions such as frequent washing, especially washing with harsh products, lack of hygiene, trauma, decreased peripheral satisfaction, immobility, incontinence, diabetes, vascular changes, malnutrition, use of multiple medications, depression, and dementia are. Among the situations that increase the risk of deterioration in skin health. For these reasons, skin care and protecting the integrity of the skin are the main goals of acute and long-term care. Physiological and pathological skin changes occur in the elderly: aged skin contains less collagen elastin and fatty tissue; skin elasticity decreases and shrinkage of the subcutaneous tissue occurs, resulting in the appearance of wrinkles and folds; the skin also has a decreased sebaceous gland and sweat gland activity causes the skin to become dry (xerosis) and more fragile; Arteriosclerotic changes in small and large vessels lead to thinning of the vessel walls and reduced blood flow to the extremities and therefore skin microcirculation.In this study; A protocol that protects the skin health of elderly patients was developed and a randomized controlled experiment was conducted to determine the effect of this protocol on skin moisture, dermatological quality of life and patient comfort in elderly patients. This thesis study is a randomized controlled experimental study with experimental and control groups and three follow-ups. In a similar study in the relevant literature, the effect size for skin moisture difference was calculated as 1.25 in the study conducted by Milani and Sparavigna (2017). In order to exceed the 95% value in determining the power of the study; 36 people, 18 in the groups, should be reached at a significance level of 5% and an effect size of 1.25 (df=34; t=2.032). In the study, it was aimed to reach a total of 44 people, 22 in the groups, considering the high power of the test and the losses.Patient Information Form, Dermatological Quality of Life Index, General Comfort Scale, Elderly Patient's Skin Evaluation Subjective Data Form, Elderly Patient's Skin Evaluation Objective Data Form, Elderly Patient's Pressure Injury Evaluation Form, Skin Moisture Measurement (DMM Skin Moisture Meter Device) will be used. Research data will be evaluated with the SPSS package program. Statistical significance level will be accepted as p<0.005 and p<0.001. CONSORT 2018 flow diagram was used in the study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are over 60 years of age, able to communicate, have not taken a bath in the last 24 hours, have not used skin moisture care products, and have not undergone any surgery in the last 6 months who voluntarily participate in the study will be included in the study (Hannel et al. 2017, Matsumoto et al. 2019, Cowdell et al. 2020).

Exclusion Criteria:

* Patients with extreme pain who receive radiotherapy chemotherapy, are allergic to any cleaning agent, and do not volunteer to participate in the study (Konya et al. 2021). He/she will be excluded from the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-05-13 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Patient Information Form (PIF) | one week
  The patient information form (PIF) was created by the researcher by scanning the literature on the subject (Bickley et al. 2017, Güner et al. 2017, Tarakçıoğlu Çelik 2019, Kalaycı and Özkul 2019, Dinçer and Kurşun 2019, İn and Akça 2021, Çelenk and Kumcağız 2022, Bekircan and Okanlı 2023).
General Comfort Scale (GCS): | one week
  Kolcaba developed the General Comfort Scale (GCS) and published it in 1992. Its Turkish validity and reliability were tested by Kuğuoğlu and Karabacak in 2008. For convenience, the four-point Likert type is mostly used. Subdimensions of the scale; relief (16 items), relaxation (17 items) and overcoming problems (15 items). Positive and negative items are given mixed in the scale. In positive questions, 4 points indicate high comfort and 1 point indicates low comfort. In negative questions, 1 point indicates high comfort and 4 points indicate low comfort. When calculating the score from the scale, negative scores are reverse coded and summed with positive items. The highest score of the scale is 192 and the lowest score is 48. Cronbach's alpha value of the Turkish version of the scale is 0.85.
Dermatological Quality of Life index (DLQI) | one week
  The scale was developed by Finlay and Khan in 1994. Turkish validity and reliability were determined by Öztürkcan et al. (2006). There are 10 questions in total, the score varies between 0-30, and there is an inverse relationship between the score obtained and quality of life. It is attempted to determine to what extent the disease-specific symptoms affect people in the last week (Namdar and Arıkan 2019). Scoring is as follows: "quite a lot = 3 points", "a lot = 2 points", "slightly = 1 point", "not at all = 0 points" and "not relevant = 0 points", and the scale can vary between 0 and 30 by adding the points of each question. The total score is obtained.
Elderly Patient's Skin Evaluation Subjective Data Form(EPSESDF) | one week
  The form was reviewed by scanning the literature (Weber and Kelley 2014, Lynn 2015, Bickley et al. 2017, Şendir and Büyükyılmaz 2017, Karadakovan 2017, Bayraktar and Faydalı 2017, Jarvis and Eckhardt 2020, Berman et al. 2021, Demir Dikmen 2021) and "Leather Care Prepared in accordance with the protocol
Elderly Patient's Skin Evaluation Objective Data Form (EPSEODF) | one week
  The form was created in line with the relevant literature (Weber and Kelley 2014, Lynn 2015, Bickley et al. 2017, Şendir and Büyükyılmaz 2017, Çatıker 2018, Jarvis and Eckhardt 2020).
Elderly Patient's Pressure Injury Evaluation Form (EPPIEF) | one week
  Form-related literature (Şendir and Büyükyılmaz 2017, EPUAP/NPIAP/PPPIA 2019, Jarvis and Eckhardt 2020, Ersoy et al. 2018, Şendir et al. 2021, Horasan 2021, https://sbn.saglik.gov.tr/BKindeksi Access It was created in accordance with the date: 1.01.2024).
Elderly Patient's Skin Care and Hygiene Evaluation Forms (EPSCHEF) | one week
  The form was prepared in line with the relevant literature (Zaybak A, Güneş 2009, Uğur 2018, Jarvis and Eckhardt 2020, Berman et al. 2021, İn and Akça 2021, Potter et al. 2021).
Skin Moisture Measurement (DMM) | one week
  To evaluate skin moisture, measurements were made with the DMM skin moisture meter. The DMM device measures moisture in any part of the skin. The amount of moisture is measured from the outer surface of this device without causing any damage.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu AKÇA, Principal Investigator — Kafkas University, Faculty of Health Sciences; Arzu KARABAĞ AYDIN, Study Director — Kafkas University, Faculty of Health Sciences
Locations (1):
- Kafkas University, Faculty of Health Sciences, Kars, Turkey/Kars, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brooks J, Cowdell F, Ersser SJ, Gardiner ED. Skin cleansing and emolliating for older people: A quasi-experimental pilot study. Int J Older People Nurs. 2017 Sep;12(3). doi: 10.1111/opn.12145. Epub 2017 Jan 12. PMID 28078772
- [Background] Konya I, Iwata H, Hayashi M, Akita T, Homma Y, Yoshida H, Yano R. Effectiveness of weak wiping pressure during bed baths in hospitalized older adults: A single-blind randomized crossover trial. Geriatr Nurs. 2021 Nov-Dec;42(6):1379-1387. doi: 10.1016/j.gerinurse.2021.09.008. Epub 2021 Sep 25. PMID 34583237
- [Background] Hahnel E, Blume-Peytavi U, Trojahn C, Dobos G, Jahnke I, Kanti V, Richter C, Lichterfeld-Kottner A, Garcia Bartels N, Kottner J. Prevalence and associated factors of skin diseases in aged nursing home residents: a multicentre prevalence study. BMJ Open. 2017 Sep 24;7(9):e018283. doi: 10.1136/bmjopen-2017-018283. PMID 28947467
- [Background] Shishido I, Yano R. Pilot study on benefits of applying a hot towel for 10 s to the skin of elderly nursing home residents during bed baths: Towards safe and comfortable bed baths. Geriatr Nurs. 2017 Sep-Oct;38(5):442-447. doi: 10.1016/j.gerinurse.2017.02.008. Epub 2017 Mar 31. PMID 28366230
- [Background] Serra R, Ielapi N, Barbetta A, de Franciscis S. Skin tears and risk factors assessment: a systematic review on evidence-based medicine. Int Wound J. 2018 Feb;15(1):38-42. doi: 10.1111/iwj.12815. Epub 2017 Oct 17. PMID 29045078
- [Background] Cowdell F, Jadotte YT, Ersser SJ, Danby S, Lawton S, Roberts A, Dyson J. Hygiene and emollient interventions for maintaining skin integrity in older people in hospital and residential care settings. Cochrane Database Syst Rev. 2020 Jan 23;1(1):CD011377. doi: 10.1002/14651858.CD011377.pub2. PMID 32006460
- [Background] Matsumoto C, Nanke K, Furumura S, Arimatsu M, Fukuyama M, Maeda H. Effects of disposable bath and towel bath on the transition of resident skin bacteria, water content of the stratum corneum, and relaxation. Am J Infect Control. 2019 Jul;47(7):811-815. doi: 10.1016/j.ajic.2018.12.008. Epub 2019 Jan 10. PMID 30639096
- [Background] Lichterfeld-Kottner A, El Genedy M, Lahmann N, Blume-Peytavi U, Buscher A, Kottner J. Maintaining skin integrity in the aged: A systematic review. Int J Nurs Stud. 2020 Mar;103:103509. doi: 10.1016/j.ijnurstu.2019.103509. Epub 2019 Dec 23. PMID 31945604